CLINICAL TRIAL: NCT00421785
Title: Effect of N-Acetylcysteine on Peritoneal Membrane Function in Chronic Peritoneal Dialysis Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 346147CTIL
Record Dates: First submitted 2007-01-11; First posted 2007-01-12 (Estimated); Last update posted 2007-07-09 (Estimated); Status verified 2007-07

CONDITIONS: ESRD; Peritoneal Dialysis
Keywords: N-acetylcysteine; Peritoneal Dialysis; ADMA
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Acetylcysteine

INTERVENTIONS:
Drug: Oral N-Acetylcysteine 1200 mg x 2/day for 4 weeks.

SUMMARY:
The aim of our study is to investigate the effect of N-acetylcysteine on peritoneal small solute clearance and removal of salt and water in prevalent CAPD patients.

DETAILED DESCRIPTION:
Cardiovascular disease is the commonest cause of morbidity and mortality in chronic dialysis patients, including those treated with CAPD (Continuous Ambulatory Peritoneal Dialysis) [1]. Uncontrolled arterial hypertension in ESRF leads to progression of LVH, which is a strong predictor for coronary events, CHF and mortality [2]. Fluid overload is a major factor in the pathogenesis of arterial hypertension in CAPD patients [3]. Therefore, interventions to optimize volume status, and hence blood pressure, are considered central in the management of such patients. Such therapies include restricting dietary sodium and water intake, use of diuretics in patients with residual renal function and optimization of peritoneal ultrafiltration with sodium and water removal [1]. As shown in the EAPOS Study, peritoneal ultrafiltration was important predictor of mortality [4].

Peritoneal fluid and salt removal can be increased by using a more hypertonic dialysis fluid using glucose as osmotic agent. Consistent use of hypertonic glucose solutions may damage peritoneal membrane and may also lead to increased systemic absorption of glucose with subsequent hyperglycemia, increased thirst and excessive water drinking. Concerns about the role of glucose in deterioration of peritoneal membrane function have been supported in recent studies [5]. Generally, the evolution of peritoneal membrane properties over time is characterized by a progressive increase in small solute transport, leading to higher glucose absorption rate from peritoneal fluid and loss of ultrafiltration capacity [6]. Such a high peritoneal transport status is associated with less peritoneal fluid removal, overhydration, hypertension and LVH. High peritoneal transport status is a risk factor of mortality in CAPD patients [7].

In recent years, there has been an increasing focus on association between inflammation, increased oxidative stress and high peritoneal transport rate and their relation to mortality in CAPD patients [8 ]. Inflammation has been shown to increase a peritoneal transport rate in CAPD patients [8]. Both inflammation and increased oxidative stress may impact to inadequate fluid removal. The exact mechanism of this phenomenon is not fully understood.

Several experimental and clinical studies showed that increased oxidative stress in dialysis patients may be due to inhibition of nitric oxide (NO) synthesis by ADMA (Asymmetric Dimethylarginine ), known to be endogenous inhibitor of NO synthetase [9]. ADMA may be significantly reduced by dialysis [10]. Metabolism of ADMA is primarily by the enzyme DDAH , which activity is decreased by inflammation, oxidative stress, diabetes mellitus and hypercholesterolemia [11]. It was proposed that circulating ADMA may be one mechanism accounting for the resistant hypertension and fluid overload in dialysis patients [11].

Based on current knowledge, treatment aimed at reducing oxidative stress should decrease ADMA levels [11], and it is logical to suggest that such a therapy might improve BP control and fluid status in CAPD patients. In our opinion, it is worth to check an ability of antioxidant therapy to produce a favorable effect on biological properties of peritoneal membrane. One preliminary study on effect of antioxidant Vitamin E showed a small beneficial effect on ADMA in chronic kidney disease [12].

N-Acetylcysteine (NAC) is an active antioxidant proved to be safe and beneficial in hemodialysis patents [13]. In our recent study, NAC effectively reduced the ototoxic effect of gentamicin in chronic hemodialysis patients [14].

The aim of our study is to investigate the effect of N-acetylcysteine on peritoneal small solute clearance and removal of salt and water in prevalent CAPD patients.

ELIGIBILITY:
Inclusion Criteria:

* The study will include 20 patients with ESRD, treated with chronic peritoneal dialysis .

Exclusion Criteria:

* Recently started treated with chronic dialysis: less than 3 months.
* Survived recent peritonitis in the last 3 months.
* Patients with acute renal failure
* Currently treated with antioxidants ( NAC, vitamin E ets.)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-02; Study Completion 2008-01 (Estimated)

PRIMARY OUTCOMES:
dualysis adequacy | 1 month
Change in peritoneal small solute transport, measured as adequacy of urea removal - Kt/V.
Change in peritoneal ultrafiltration rate on PET test.

SECONDARY OUTCOMES:
Change in residual kidney function
Change in Body Weight and Blood Pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Leonid S Feldman, MD, Principal Investigator — Assaf Harofeh MC
Locations (1):
- Dialyss unit, Ẕerifin, Israel